CLINICAL TRIAL: NCT02973854
Title: Activation of the Sphingosine-1-phosphate (S1P) to S1P1 Receptor Subtype (S1PR1) Axis in Patients With Endometriosis: Identification of Potential Relevant Biomarkers to Diagnose and Treat
Acronym: S1P1
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Patrick Yeung Jr., MD, MD, St. Louis University
Other Study IDs: 25996
Record Dates: First submitted 2016-10-04; First posted 2016-11-25 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Per the PI's standard surgical approach to endometriosis, all areas of abnormal peritoneum will be excised (removed).
  After surgical excision has been performed, in order to provide standardized specimens for our research, a 3mm punch biopsy will be obtained from the excised peritoneum tissue. The 3 mm biopsy will be sent for research analysis, and the rest of the excised peritoneum tissue will be sent to histology (SSM) for evaluation and classification as having endometriosis or not. For each patient in the study, blood will also be collected to look for markers for endometriosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients seen at the SLUCare Center for Endometriosis (including those with or without pain) undergoing laser excision surgery for known or suspected endometriosis will be recruited for the study.

Per the PI's standard surgical approach to endometriosis, all areas of abnormal peritoneum will be excised (removed).

After surgical excision has been performed, in order to provide standardized specimens for our research, a 3mm punch biopsy will be obtained from the excised peritoneum tissue. The 3 mm biopsy will be sent for research analysis, and the rest of the excised peritoneum tissue will be sent to histology (SSM) for evaluation and classification as having endometriosis or not. For each patient in the study, blood will also be collected to look for markers for endometriosis.

DETAILED DESCRIPTION:
The study is investigator-initiated, prospective, comparative study. Laparoscopic surgery for endometriosis on patients presenting with pain, infertility or both will be performed by the principal investigator at St. Mary's Hospital. We will be collecting preoperative, operative and postoperative follow-up data on all patients recruited for this study based on comprehensive preoperative questionnaires, which includes data collection on pain scores (by VAS scales) and standardized QOL scales, and the 6-12 month follow questionnaire. The surgical approach in the treatment of endometriosis is by excision only, so that all lesions (abnormal areas of peritoneum) are excised resulting in tissue specimens that are classified at a histologic level, which is the gold standard way to diagnose the presence of endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen at the Center for Endometriosis (including those with or without pain) who are undergoing excision surgery.
* Patients who are undergoing laser excision surgery for known or suspected endometriosis will be recruited for the study.
* Completed a preoperative questionnaire

Exclusion Criteria:

* prior bilateral salpingo-oophorectomy
* post natural menopause

Ages: 13 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients seen at the Center for Endometriosis (including those with or without pain) undergoing laser excision surgery for known or suspected endometriosis will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
S1PR1 levels in PBLs with and without endometriosis. | At Surgery
  To determine if S1PR1 levels in PBLs can discriminate between patients with endometriosis and patients without endometriosis.

CONTACTS AND LOCATIONS:
Locations (1):
- SSM St. Mary's, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No